CLINICAL TRIAL: NCT04621422
Title: Contribution of New Generation Oxford Nanopore-type High-throughput Sequencing in the Diagnostic Strategy of Neurogenetic Diseases.
Acronym: NEURONGS3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/51
Record Dates: First submitted 2020-10-12; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Neuro-Degenerative Disease
MeSH Terms: interventions — Myotonin-Protein Kinase; CNBP protein, human; Lipoproteins, HDL2; Frataxin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 5 to 10 µg of DNA samples per patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Subject carrying an amplification of nucleotide repeats in one of the following 9 genes FMR1, DMPK, ZNF9, SCA2, JPH3, HD, FXN, C9ORF72, RFC1 — Biological/Vaccine: DNA Samples collection as part of usual care

SUMMARY:
Since 2012, NGS sequencing of long fragments or long reads has developed in various fields of research and today presents itself as a very promising alternative solution in the analysis of repeat amplifications. The Oxford Nanopore NGS automaton offers the prospect of bringing together 1st and 2nd line analyzes of all loci potentially indicated in neurogenetics at the same time. The project aims to compare the use of this new technology with methods currently used in reference laboratories.

The main objective is to evaluate the ability of next-generation high-throughput Oxford Nanopore-type sequencing (NEURONGS3) to diagnose 9 neurogenetic diseases compared to reference protocols via PCR (+/- Southern blot).

The secondary objective is to evaluate the repeatability of the NGS (intra-sample reproducibility) analysis in the diagnosis of 8 neurogenetic diseases.

DETAILED DESCRIPTION:
Since 2012, NGS sequencing of long fragments or long reads has developed in various fields of research and today presents itself as a very promising alternative solution in the analysis of repeat amplifications. The Oxford Nanopore NGS automaton offers the prospect of bringing together 1st and 2nd line analyzes of all loci potentially indicated in neurogenetics at the same time. The project aims to compare the use of this new technology with methods currently used in reference laboratories.

Multicenter cross-sectional early phase diagnostic study on already existing biological collections. Analyzes with the new technique (NGS) will be carried out blinded to the results obtained with the current reference algorithm based on the sequential performance of PCRs The main objective is to evaluate the ability of next-generation high-throughput Oxford Nanopore-type sequencing (NEURONGS3) to diagnose 9 neurogenetic diseases compared to reference protocols via PCR (+/- Southern blot).

The secondary objective is to evaluate the repeatability of the NGS (intra-sample reproducibility) analysis in the diagnosis of 8 neurogenetic diseases.

ELIGIBILITY:
Inclusion Criteria:

* minors, adults and protected adults.
* Subject carrying an amplification of nucleotide repeats in one of the following 9 genes FMR1, DMPK, ZNF9, SCA2, JPH3, HD, FXN, C9ORF72, RFC1
* DNA available in sufficient quantity (5 to 10 µg)

Exclusion Criteria:

* DNA degraded or of medium size <30kb,
* Patient objection to research - This patient objection must be reached to the center's investigator within 1 maximum period of 1 month after sending the information note.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject carrying an amplification of nucleotide repeats in one of the following 9 genes FMR1, DMPK, ZNF9, SCA2, JPH3, HD, FXN, C9ORF72, RFC1
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients tested positive by Next Generation Sequencing among all the patients tested positive by the current algorithm based on PCRs | through study completion, an average of 2 years
  For each of the 9 considered diseases, the proportion will be established as well as its 95% confidence interval.

SECONDARY OUTCOMES:
Difference between the number of repetition amplifications found by the Next Generation Sequencing method and the number of repetition amplifications found by the PCR diagnosis method | through study completion, an average of 2 years
  For each of the 9 considered diseases, the number of repetition amplifications found by the Next Generation Sequencing method will be compared to the number of repetition amplifications found by the PCR diagnosis method using the Bland et Altman graphs. The average and standard deviation of the difference will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Goizet, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No